CLINICAL TRIAL: NCT00842465
Title: Characterization and Implication of Prolactin Receptor Mutants in Human Breast Diseases
Brief Title: Prolactin Receptor and Breast Diseases
Acronym: Prolacsein
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: P070608
Record Dates: First submitted 2009-01-13; First posted 2009-02-12 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-10

CONDITIONS: Benign Breast Disease; Breast Cancer
Keywords: Breast diseases,; human mutation,; prolactin receptor;; breast cancer
MeSH Terms: conditions — Cystic Fibrosis; Breast Neoplasms; Breast Diseases | interventions — Surgical Procedures, Operative; Blood Specimen Collection; High-Energy Shock Waves; Bone Density

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood collection breast Biopsy or surgery
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: benign breast diseases
  Interventions: Biological: blood collection for hormonal status analysis; Procedure: breast Biopsy or surgery; Genetic: blood collection; Other: ultrasonography (pelvis and breast), bone mineral density
- 2: breast cancer
  Interventions: Biological: blood collection for hormonal status analysis; Procedure: breast Biopsy or surgery; Genetic: blood collection; Other: ultrasonography (pelvis and breast), bone mineral density
- 3: control
  Interventions: Biological: blood collection for hormonal status analysis; Genetic: blood collection

INTERVENTIONS:
Biological: blood collection for hormonal status analysis — for hormonal status analysis
Procedure: breast Biopsy or surgery — breast Biopsy or surgery
  Groups: 1; 2
Genetic: blood collection — blood collection for prlR gene sequencing
Other: ultrasonography (pelvis and breast), bone mineral density — ultrasonography (pelvis and breast), bone mineral density
  Groups: 1; 2

SUMMARY:
Prolactin is known to play an important role in breast development and differentiation. Thus proliferative breast diseases are good models to unravel PRl / PRLR function in proliferative processes.

The aim of this project is to identify and to characterize new mutants of the prolactin receptor gene within cohorts of benign or malign breast diseases with low or high occurrence frequency in human populations

DETAILED DESCRIPTION:
There is currently no known genetic disease linked to prolactin (prl) or its receptor (prlR) in humans. In a previous work, we have identified a new mutation of prolactin receptor that leads to it's constitutive activation and to cell proliferation signalling cascades (i.e. through MAP kinases).

This result suggests that PRLR mutants may have a strong physiopathological impact on breast diseases etiology and/or development and/or evolution.

Based on this, we will pursue the identification of new PRLR mutants in various breast diseases and continue their in vitro functional characterization and then analyse their in vivo consequences on breast tissue samples collected within these women.

1. In a first time we wish to confirm our previous results on multiple fibroadenomas (MFA). The current cohort will be augmented with 30 to 35 new patients each year. We will confirm our in vitro results in vivo with tumoral and peri-tumoral tissue samples.
2. We then wish to extend this study to other rare breast pathologies (i.e. gigantomastia, phyllodies tumors, giant fibroadenomas) and to more common ones (simple fibroadenomas) to demonstrate a link between simple FA and MFA.
3. in a third time we will try to determinate whether a constitutive activation of PRLR leads to enhanced occurrence of benign / malign transitions.

ELIGIBILITY:
Inclusion criteria :

* benign breast diseases

  * 10 < age < 25 for simple FA
  * 10 < age < 50 for other diseases .no hormonal treatment for at least 3 months if patients took cyproterone acetate; 1 month for other ovaries-interfering hormonal treatment, and 1 week for ovaries-non-interfering hormonal treatments.
  * Signature of the informed consent form (icf) by patients or their legal representative (for patients under age of 18.)
* breast cancer :

  * having a breast cancer with a planned surgery
  * age > 55 years
  * post menopausal with not menopause substitution treatment
  * signature of the icf
* control group :

  * 18 < age < 60
  * signature of the icf

Exclusion criteria :

* no signature or no conformity of the icf
* no social security

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Benign breast diseases(60 simple FA, 71 other breast diseases) Brest Cancer : 132 Control : 525
Sampling Method: Non-Probability Sample
Enrollment: 735 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Sequencing of PRLR | at inclusion

SECONDARY OUTCOMES:
Breast ultrasonography | at inclusion
Breast MRI | at inclusion
Pelvic ultrasonography | at inclusion
Bone mineral density measurement | at inclusion
Hormonal and metabolic evaluation | at inclusion
Histological analysis of tumoral and peri-tumoral tissues | at surgery
Tumor transcriptome analysis | at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Touraine, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France